CLINICAL TRIAL: NCT02284386
Title: Evaluation of the Pharmacokinetics and Safety of Bupivacaine HCl Spinal Block and EXPAREL Local Infiltration in Subjects Undergoing for Unilateral Total Knee Arthroplasty
Brief Title: Pharmacokinetics and Safety of Bupivacaine HCl Spinal Block and EXPAREL Local Infiltration in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-405
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Pain
Keywords: Total knee arthroplasty
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupivacaine SNB + EXPAREL Infiltration (Experimental): Spinal block with bupivacaine HCl 7.5 mg/mL. Local infiltration of EXPAREL 266 mg.
  Interventions: Drug: Bupivacaine SNB; Drug: EXPAREL Infiltration

INTERVENTIONS:
Drug: Bupivacaine SNB — SNB with a single 1.6 mL dose of bupivacaine HCl 7.5 mg/mL within 2 hours prior to the surgical procedure.
  Other Names: Bupivacaine
Drug: EXPAREL Infiltration — Local infiltration of EXPAREL 266 mg into the surgical site at the end of the surgery just prior to wound closure.
  Other Names: Bupivacaine

SUMMARY:
This is a Phase 4, multicenter, open-label study designed to characterize the pharmacokinetic (PK) profile of total bupivacaine in approximately 15 adult subjects undergoing primary unilateral total knee arthroplasty (TKA) with bupivacaine hydrochloride (HCl) spinal nerve block (SNB) and EXPAREL local infiltration into the surgical site.

DETAILED DESCRIPTION:
On Day 1, following an epinephrine "wash" of the spinal block syringe, eligible subjects will receive a single 1.6 mL dose of bupivacaine HCl 7.5 mg/mL within 2 hours prior to the surgical procedure as a spinal block. EXPAREL 266 mg in 20 mL (expanded with 70 mL of preservative-free sterile normal saline to a total volume of 90 mL) will be infiltrated into the surgical site at the end of the surgery prior to wound closure. There will be no local co-administration of the two drugs.

Blood samples for bupivacaine PK analysis will be obtained from subjects at baseline (prior to bupivacaine HCl administration for nerve block), 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 48, and 72 hours after the beginning of EXPAREL administration, and on Day 14.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age.
2. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
3. Scheduled to undergo spinal block in conjunction with unilateral TKA.
4. Female subjects must be surgically sterile, at least 2 years postmenopausal, or using a medically acceptable method of birth control. Females of childbearing potential must have a documented negative blood or urine pregnancy test result within 24 hours before surgery.
5. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.

Exclusion Criteria:

1. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics or opioids.
2. Contraindication to bupivacaine.
3. Received bupivacaine or any other local anesthetic within 7 days of EXPAREL administration.
4. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after EXPAREL administration.
5. Planned concurrent surgical procedure (e.g., bilateral TKA).
6. Body weight <50 kg (110 pounds) or a body mass index ≥45 kg/m2.
7. Received any investigational drug within 30 days prior to EXPAREL administration, and/or has planned administration of another investigational product or procedure during the subject's participation in this study.
8. Previous participation in an EXPAREL study.
9. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
10. Current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postsurgical course.
11. Clinically significant medical or psychiatric disease that, in the opinion of the Investigator, would constitute a contraindication to participation in the study, or cause inability to comply with the study requirements.

    In addition, the subject will be ineligible to receive EXPAREL if he or she meets the following criteria during surgery:
12. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hutchins, MD, Principal Investigator — University of Minnesoty
Locations (2):
- United States (2):
  - Shaols Medical Trials, Inc., Sheffield, Alabama
  - University of Minnesota Medical Center - Fairview, West Bank, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing total knee arthroplasty
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 67.8 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: baseline, 15,30 min, 1,2,4,8,12,24,48,72 hours post dose, day 14
Population: Of 15 subjects, one subject was removed as an outlier
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Number analyzed (Participants) | 14
ng/mL | 408 (161)

2. Primary Outcome: Time to Peak Plasma Concentration (Tmax)
Time Frame: baseline, 15,30 min, 1,2,4,8,12,24,48,72 hours post dose, day 14
Measure: Median (Full Range); unit: hours
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Number analyzed (Participants) | 15
hours | 12.0 [0.47 to 52.5]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Collection Time After Drug Administration (AUC0-last)
Time Frame: baseline, 15,30 min, 1,2,4,8,12,24,48,72 hours post dose, day 14
Measure: Mean (Standard Deviation); unit: hours x ng/mL
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Number analyzed (Participants) | 14
hours x ng/mL | 15286 (8017)

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity After Drug Administration (AUC0-∞)
Time Frame: baseline, 15,30 min, 1,2,4,8,12,24,48,72 hours post dose, day 14
Measure: Mean (Standard Deviation); unit: hours x ng/mL
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Number analyzed (Participants) | 10
hours x ng/mL | 13741 (4627)

5. Primary Outcome: The Apparent Terminal Elimination Rate Constant (λz)
Time Frame: baseline, 15,30 min, 1,2,4,8,12,24,48,72 hours post dose, day 14
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Number analyzed (Participants) | 10
1/hours | 0.0523 (0.0164)

6. Primary Outcome: The Apparent Terminal Elimination Half-life (t1/2el)
Time Frame: baseline, 15,30 min, 1,2,4,8,12,24,48,72 hours post dose, day 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Number analyzed (Participants) | 10
hours | 14.7 (5.44)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Bupivacaine SNB + EXPAREL Infiltration
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 12/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine SNB + EXPAREL Infiltration (N=15)
Nausea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 2
Anaemia Postoperative (Injury, poisoning and procedural complications) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Blood Pressure Increased (Investigations) | 1
Body Temperature Increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No